CLINICAL TRIAL: NCT04170192
Title: Multi-center Clinical Study of Cord Blood Stem Cell Transplantation in The Treatment of Very Early-Onset Inflammatory Bowel Disease Caused by Interleukin-10 Receptor Gene Deficiency
Brief Title: Multi-center Clinical Study of Cord Blood Stem Cell Transplantation for IBD Caused by IL-10R Gene Deficiency
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Hospital (Other); Children's Hospital of Soochow University (Other); Beijing Children's Hospital (Other); Guangzhou Women and Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); Wuhan Women and Children's Medical Center (Other); Children's Hospital of Nanjing Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Xiaowen Zhai, vice president, Children's Hospital of Fudan University
Other Study IDs: CPBMT-IBD-2019
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Umbilical Cord Blood Stem Cell Transplantation; Inflammatory Bowel Disease; Interleukin 10 Receptor
MeSH Terms: conditions — Inflammatory Bowel Diseases; Inflammatory Bowel Disease 28, Autosomal Recessive | interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample of every patient will be collected pre and post-transplant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UCBT-IBD-Case: Very early onset IBD patients who underwent Cord Blood Stem Cell Transplantation.
  Interventions: Procedure: Cord Blood Stem Cell Transplantation

INTERVENTIONS:
Procedure: Cord Blood Stem Cell Transplantation — Unrelated cord blood stem cell selection; Reduced intensity conditioning regime; GVHD prevention; Infection prevention.

SUMMARY:
Very early onset inflammatory bowel disease (VEO-IBD) is a special subtype of children's inflammatory bowel disease (IBD). VEO-IBD is mostly caused by single-gene defects and can be cured by allo-hematopoietic stem cell transplantation ( HSCT). Umbilical Cord Blood Transplantation (UCBT) is less reported in these patients.

DETAILED DESCRIPTION:
Very early onset inflammatory bowel disease (VEO-IBD) is a special subtype of children's inflammatory bowel disease (IBD). The clinical characteristics of VEO-IBD patients include early onset, severe diarrhea, severe malnutrition, perianal diseases and repeated infection. Studies have found that VEO-IBD is mostly caused by single-gene defects and can be cured by allo-hematopoietic stem cell transplantation ( HSCT). VEO-IBD is a rare disease. At present, there is no large sample of clinical data for transplantation in these patients. Umbilical Cord Blood Transplantation (UCBT) is less reported. Therefore, many transplantation-related issues need to be further studied, including HSCT indications, transplantation timing, pre-transplantation drug therapy, intestinal protection during transplantation, prevention and treatment of post-transplantation complications and so on. The aim of this study is to investigate the efficacy of UCBT in the treatment of VEO-IBD caused by interleukin-10 receptor (IL10R) gene deficiency, including engraftment rate, disease-free survival rate and overall survival rate, and to evaluate transplant-related mortality and complications. All the selected cases are diagnosed as VEO-IBD with IL10R gene deficiency by enteroscopy, histopathology and gene detection. These patients have no matched sibling donors. Their organs function should be normal. The guardian of the patient has the desire and requirement for UCBT and signs the informed consent before treatment. Cord blood stem cell selection: HLA high-resolution detection of patients before transplantation, searching through cord blood stem cell bank, selecting cord blood stem cells that meet the following criteria: HLA-A, B, C, DRB1 high-resolution (genotype) > 6/8 matching, total number of nuclear cells > 5 x 10^7/kg. Conditioning regimen: fludarabine + busulfan + cyclophosphamide. GVHD prevention: tacrolimus (FK506) or cyclosporine A. Infection prevention: Micafungin/caspofungin before engraftment, voriconazole after engraftment to prevent fungi. Ganciclovir is used from the beginning of conditioning to the infusion of cord blood stem cells, and acyclovir is used to prevent virus infection. SMZ is used to prevent Pneumocystis carinii infection after engraftment until half a year after the withdrawal of immunosuppressive agents.

Procedure/Surgery: Cord Blood Stem Cell Transplantation Unrelated cord blood stem cell selection: HLA high-resolution detection should be performed before transplantation. High-resolution (genotype) matching of HLA-A, B, C and DRB1 should be selected. The total number of nuclear cells should be more than 5*107/kg.

Conditioning regime: fludarabine 30 mg/m2/d for 5 days, busulfan 1 mg/kg for 4 times for 3 days, cyclophosphamide 50 mg/kg for 2 days.

Prevention of GVHD: tacrolimus (FK506) 0.1 mg/kg/day, starting from day 4 before transplantation, taking orally twice on an empty stomach to monitor the blood concentration and keep it at 5-10 ng/ml.

Infection prevention: Micafungin/caspofungin before engraftment, voriconazole after engraftment to prevent fungi. Ganciclovir is used from the beginning of conditioning to the beginning of reinfusion, and acyclovir is used to prevent virus infection until immunosuppressive agents are discontinued after reinfusion. SMZ is used to prevents Pneumocystis carinii infection after engraftment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: All selected cases will be diagnosed as very early-onset inflammatory bowel disease with interleukin-10 receptor gene deficiency through gastroenterology, pathology and gene diagnosis institutions to improve enteroscopy, histopathology and gene detection.
2. The patients have no HLA matched sibling donor.
3. All organs function normally and meet the following test criteria:

   Liver function ALT, AST < 10 times normal value upper limit, TBIL < 5 times normal value upper limit.

   Renal function BUN and Cr < 1.25 times the upper limit of normal value. ECG and echocardiography showed no cardiac insufficiency.
4. The legal guardian of the patient has the desire and requirement for the treatment of allogeneic umbilical cord blood stem cell transplantation, and signs the informed consent before treatment. The informed consent should inform all relevant contents of clinical research, patients are willing and abide by the treatment plan, follow-up plan, laboratory examination, etc.

Exclusion Criteria:

1. There are any contraindications of hematopoietic stem cell transplantation.
2. There are other serious diseases, such as severe damage to vital organ functions: respiratory failure, cardiac insufficiency, decompensated liver insufficiency, renal insufficiency, uncontrollable infection and so on.
3. Other drug clinical researchers are under way.
4. Simultaneously suffering from other serious acute or chronic physical or mental diseases, or abnormal laboratory examinations, may affect patient's life safety and compliance, and affect informed consent, research participation, follow-up or result interpretation.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with very early-onset inflammatory bowel disease with interleukin-10 receptor gene deficiency through gastroenterology, pathology and gene diagnosis institutions to improve enteroscopy, histopathology and gene detection.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 3 years after transplantation
  Overall survival is defined as the survival status of patients by the end of 3 years after the transplanting, coded as 1 for dead and 0 for survive.

SECONDARY OUTCOMES:
Disease free survival rate | 3 years after transplantation
  Disease free survival is defined as the survival status of patients by the end of the third year after transplantation. Disease free survival is defined as survive without conditions including engraftment failure and death caused by any reasons. The variable is coded as 0 for disease free survive, and 1 for all conditions other than the defined status of "0".
Successful engraftment | 3 years after transplantation
  The event of successful engraftment is defined as Neutrophil count ≥ 0.5×10^9/L for continuous 3 days and platelet count ≥ 20×10^9/L for continuous 7 days without transfusion. It is coded as 1.

OTHER OUTCOMES:
The occurrence of adverse events (AE) | 3 years after transplantation
  The adverse events (AE) is a composite variable including liver and kidney function damage, nausea, vomiting, arrhythmia and dyspnea. The variable would be coded as 1 if any of these events occurs after transplantation for 3 years while 0 for none . These adverse events would be measured by assessment scale method according to NCI CTC AE v4.0 classification standard.
The occurrence of graft-versus-host disease (GVHD) | 3 years after transplantation
  Acute and chronic GVHD is measured and graded as per standardised criteria.
Transplant-related mortality | 3 years after transplantation
  Transplant-related mortality (TRM) is defined as the proportion of non primary disease death patients in the total number of cord blood stem cell transplantation patients in the same period within 100 days after transplantation.
The occurrence of transplant-related complications except GVHD | 3 years after transplantation
  Transplant-related complications include infections, hepatic venous occlusion disease, hemorrhagic cystitis, capillary leakage syndrome, thrombotic microangiopathy, post-transplantation lymphoproliferative disease, idiopathic pneumonia syndrome and obstructive bronchiolitis, which are diagnosed according to the relevant diagnosis standards of each disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Hui, Master, Study Director — Shanghai Children's Hospital; Hu Shaoyan, PHD, Study Director — Children's Hospital of Soochow University; Qin Maoquan, PHD, Study Director — Beijing Children's Hospital; Jiang Hua, PHD, Study Director — Guangzhou Women and Children's Medical Center; Liu Sixi, Master, Study Director — Shenzhen Children's Hospital; Xiong Hao, PHD, Study Director — Wuhan Women and Children's Medical Center; Fang Yongjun, PHD, Study Director — Children's Hospital of Nanjing Medical University; Wang Dao, PHD, Study Director — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Minhang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bianco AM, Girardelli M, Tommasini A. Genetics of inflammatory bowel disease from multifactorial to monogenic forms. World J Gastroenterol. 2015 Nov 21;21(43):12296-310. doi: 10.3748/wjg.v21.i43.12296. PMID 26604638
- [Result] Kotlarz D, Beier R, Murugan D, Diestelhorst J, Jensen O, Boztug K, Pfeifer D, Kreipe H, Pfister ED, Baumann U, Puchalka J, Bohne J, Egritas O, Dalgic B, Kolho KL, Sauerbrey A, Buderus S, Gungor T, Enninger A, Koda YK, Guariso G, Weiss B, Corbacioglu S, Socha P, Uslu N, Metin A, Wahbeh GT, Husain K, Ramadan D, Al-Herz W, Grimbacher B, Sauer M, Sykora KW, Koletzko S, Klein C. Loss of interleukin-10 signaling and infantile inflammatory bowel disease: implications for diagnosis and therapy. Gastroenterology. 2012 Aug;143(2):347-55. doi: 10.1053/j.gastro.2012.04.045. Epub 2012 Apr 28. PMID 22549091
- [Result] Engelhardt KR, Shah N, Faizura-Yeop I, Kocacik Uygun DF, Frede N, Muise AM, Shteyer E, Filiz S, Chee R, Elawad M, Hartmann B, Arkwright PD, Dvorak C, Klein C, Puck JM, Grimbacher B, Glocker EO. Clinical outcome in IL-10- and IL-10 receptor-deficient patients with or without hematopoietic stem cell transplantation. J Allergy Clin Immunol. 2013 Mar;131(3):825-30. doi: 10.1016/j.jaci.2012.09.025. Epub 2012 Nov 14. PMID 23158016
- [Result] Pigneur B, Escher J, Elawad M, Lima R, Buderus S, Kierkus J, Guariso G, Canioni D, Lambot K, Talbotec C, Shah N, Begue B, Rieux-Laucat F, Goulet O, Cerf-Bensussan N, Neven B, Ruemmele FM. Phenotypic characterization of very early-onset IBD due to mutations in the IL10, IL10 receptor alpha or beta gene: a survey of the Genius Working Group. Inflamm Bowel Dis. 2013 Dec;19(13):2820-8. doi: 10.1097/01.MIB.0000435439.22484.d3. PMID 24216686
- [Result] Huang Z, Peng K, Li X, Zhao R, You J, Cheng X, Wang Z, Wang Y, Wu B, Wang H, Zeng H, Yu Z, Zheng C, Wang Y, Huang Y. Mutations in Interleukin-10 Receptor and Clinical Phenotypes in Patients with Very Early Onset Inflammatory Bowel Disease: A Chinese VEO-IBD Collaboration Group Survey. Inflamm Bowel Dis. 2017 Apr;23(4):578-590. doi: 10.1097/MIB.0000000000001058. PMID 28267044
- [Result] Silverberg MS, Satsangi J, Ahmad T, Arnott ID, Bernstein CN, Brant SR, Caprilli R, Colombel JF, Gasche C, Geboes K, Jewell DP, Karban A, Loftus EV Jr, Pena AS, Riddell RH, Sachar DB, Schreiber S, Steinhart AH, Targan SR, Vermeire S, Warren BF. Toward an integrated clinical, molecular and serological classification of inflammatory bowel disease: report of a Working Party of the 2005 Montreal World Congress of Gastroenterology. Can J Gastroenterol. 2005 Sep;19 Suppl A:5A-36A. doi: 10.1155/2005/269076. PMID 16151544
- [Result] Levine A, Griffiths A, Markowitz J, Wilson DC, Turner D, Russell RK, Fell J, Ruemmele FM, Walters T, Sherlock M, Dubinsky M, Hyams JS. Pediatric modification of the Montreal classification for inflammatory bowel disease: the Paris classification. Inflamm Bowel Dis. 2011 Jun;17(6):1314-21. doi: 10.1002/ibd.21493. Epub 2010 Nov 8. PMID 21560194
- [Result] Uhlig HH, Schwerd T, Koletzko S, Shah N, Kammermeier J, Elkadri A, Ouahed J, Wilson DC, Travis SP, Turner D, Klein C, Snapper SB, Muise AM; COLORS in IBD Study Group and NEOPICS. The diagnostic approach to monogenic very early onset inflammatory bowel disease. Gastroenterology. 2014 Nov;147(5):990-1007.e3. doi: 10.1053/j.gastro.2014.07.023. Epub 2014 Jul 21. PMID 25058236
- [Result] Kelsen JR, Dawany N, Moran CJ, Petersen BS, Sarmady M, Sasson A, Pauly-Hubbard H, Martinez A, Maurer K, Soong J, Rappaport E, Franke A, Keller A, Winter HS, Mamula P, Piccoli D, Artis D, Sonnenberg GF, Daly M, Sullivan KE, Baldassano RN, Devoto M. Exome sequencing analysis reveals variants in primary immunodeficiency genes in patients with very early onset inflammatory bowel disease. Gastroenterology. 2015 Nov;149(6):1415-24. doi: 10.1053/j.gastro.2015.07.006. Epub 2015 Jul 17. PMID 26193622
- [Result] Glocker EO, Kotlarz D, Boztug K, Gertz EM, Schaffer AA, Noyan F, Perro M, Diestelhorst J, Allroth A, Murugan D, Hatscher N, Pfeifer D, Sykora KW, Sauer M, Kreipe H, Lacher M, Nustede R, Woellner C, Baumann U, Salzer U, Koletzko S, Shah N, Segal AW, Sauerbrey A, Buderus S, Snapper SB, Grimbacher B, Klein C. Inflammatory bowel disease and mutations affecting the interleukin-10 receptor. N Engl J Med. 2009 Nov 19;361(21):2033-45. doi: 10.1056/NEJMoa0907206. Epub 2009 Nov 4. PMID 19890111
- [Result] Peng K, Qian X, Huang Z, Lu J, Wang Y, Zhou Y, Wang H, Wu B, Wang Y, Chen L, Zhai X, Huang Y. Umbilical Cord Blood Transplantation Corrects Very Early-Onset Inflammatory Bowel Disease in Chinese Patients With IL10RA-Associated Immune Deficiency. Inflamm Bowel Dis. 2018 Jun 8;24(7):1416-1427. doi: 10.1093/ibd/izy028. PMID 29788474